CLINICAL TRIAL: NCT02308319
Title: A Phase 4, Open-Label Study to Investigate the Efficacy and Safety of Tenofovir Disoproxil Fumarate (Viread(R)) in Preventing Hepatocellular Carcinoma Recurrence in Chronic Hepatitis B Virus Infected Patients With Low Viral Load at Baseline Treated With Radiofrequency Ablation or Resection
Brief Title: Prompt Or Watchful Monitoring for Hepatitis B Virus Related Hepatocellular Carcinoma Without Elevated viRal Load
Acronym: POWER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-09-149
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma, Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROMPT (Active Comparator): Prompt therapy with Tenofovir disoproxil fumarate (Viread(R)) 300mg p.o
  Interventions: Drug: Tenofovir disoproxil fumarate
- Watchful monitoring (Other): Wait and treat with Tenofovir disoproxil fumarate (Viread(R)) when active liver disease is present [defined as HBV DNA >2,000 IU/ml and abnormal ALT (>40 IU/ml)]
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — 300mg q.d. per oral
  Other Names: Viread(R)

SUMMARY:
Antiviral therapy for HBV may play an important role here, as a large observation study from Taiwan reported that the use of nucleos(t)ide analogues (NUC) was associated with 33% reduction in HCC recurrence. In the first randomized controlled trial evaluating the use of NUC after surgical resection for HCC, NUC therapy was associated with better 2-year overall (94% vs. 62%) and recurrence-free (56% vs. 20%) survival. However, patients with active liver disease should be treated regardless of their impact on HCC recurrence (patients with high serum HBV DNA and abnormal ALT). What is less clear is that whether patients with low level HBV DNA, and normal serum ALT levels should be treated to reduce HCC recurrence.

In this trial, we will investigate to determine the efficacy of the treatment with Tenofovir disoproxil fumarate (Viread(R)) as measured by the cumulative incidence rate of hepatocellular carcinoma (HCC) at 3 year after curative treatment with radiofrequency ablation (RFA) or surgical resection (SR) in chronic hepatitis B virus (HBV) infected patients with low viral load.

DETAILED DESCRIPTION:
HCC is a major global health problem, which is the third leading cause of cancer-related deaths, and accounts for 7% of all cancers worldwide. Curative treatment, such as SR, RFA has improved patients prognosis, however, even after successful curative treatment, high rates of disease recurrence limiting overall survival in HCC patients. In this regard, method to reduce HCC recurrence is an essential component of a therapeutic strategy to maximize outcome.

Antiviral therapy for HBV may play an important role here, as a large observation study from Taiwan reported that the use of NUCs was associated with 33% reduction in HCC recurrence. In the first randomized controlled trial evaluating the use of NUC after surgical resection for HCC, NUC therapy was associated with better 2-year overall (94% vs. 62%) and recurrence-free (56% vs. 20%) survival. However, patients with active liver disease should be treated regardless of their impact on HCC recurrence (patients with high serum HBV DNA and abnormal ALT). What is less clear is that whether patients with low level HBV DNA, and normal serum ALT levels should be treated to reduce HCC recurrence.

In the randomized controlled trial by Yin et al, antiviral therapy was also beneficial in Chronic hepatitis B patients with low viral load (HBV DNA < 104 copies/ml). However, there is a need for further validation of their finding for several reasons. First, the baseline characteristics between two groups were not same (more advanced tumors in the control arm). Second, the recurrence rates in the control arm was too high (about 80%), and the number of patients was small (control = 32, antiviral therapy = 22). Third, HBV DNA levels at 6 months was decreased in the antiviral therapy group (3.36 ± 0.68 log10 copies/ml vs. 4.66 ± 1.38 log10 copies/ml), but was not optimal. The used drugs were lamivudine, adefovir plus lamivudine or entecavir 0.5 mg. With more potent antiviral drug, better outcome is expected.

In this trial, we will investigate to determine the efficacy of the treatment with Tenofovir disoproxil fumarate (Viread(R)) as measured by the cumulative incidence rate of hepatocellular carcinoma (HCC) at 3 year after curative treatment with radiofrequency ablation (RFA) or surgical resection (SR) in chronic hepatitis B virus (HBV) infected patients with low viral load.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (clinically or histologically)
* chronic hepatitis B
* serum HBV DNA < 2000 IU/mL
* HCC stage BCLC 0 or A
* treated or will be treated with RFA or surgical resection

Exclusion Criteria:

* co-infected with HCV, HIV
* currently using antiviral drug (lamivudine, adefovir, clevudine, tenofovir, entecavir, telbivudine) or interferon
* other malignancy
* dialysis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
New onset ascites, variceal bleeding, hepatic encephalopathy | 3 years
Child-Pugh score and MELD score at baseline and at final follow-up | 3 years
Reactivation of hepatitis B | 3 years
  Increase in DNA 1log IU/mL at least 4 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woon Paik, M.D., Ph.D., Principal Investigator — Samsung Medical Center